CLINICAL TRIAL: NCT03086382
Title: A Randomized, Open-Label, Single-Dose, 2-Period Crossover Study to Investigate the Bioequivalence of Lacosamide Tablet (200mg) and Syrup (10mg/ml) in Healthy Chinese Male Subjects
Brief Title: A Study to Investigate the Bioequivalence of Lacosamide Tablet (200mg) and Syrup (10mg/ml) in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SP1001
Record Dates: First submitted 2017-03-20; First posted 2017-03-22 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Healthy Male Volunteers
Keywords: Lacosamide; Syrup; Bioequivalence; Tablet
MeSH Terms: interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A - B (Experimental): Single administration of Treatment A (single dose of Lacosamide (LCM) 200 mg, given as 2 tablets of LCM 100 mg under fasting conditions, followed by a Wash-Out Period of at least 7 days and a single administration of Treatment B (single dose of LCM 200 mg given as syrup) under fasting conditions
  Interventions: Drug: Lacosamide (LCM) tablet; Drug: Lacosamide (LCM) syrup
- Treatment B - A (Experimental): Single administration of Treatment B (single dose of LCM 200 mg given as syrup) under fasting conditions, followed by a Wash-Out Period of at least 7 days and a single administration of Treatment A (single dose of Lacosamide (LCM) 200 mg, given as 2 tablets of LCM 100 mg) under fasting conditions
  Interventions: Drug: Lacosamide (LCM) tablet

INTERVENTIONS:
Drug: Lacosamide (LCM) tablet — Treatment A: Single dose of Lacosamide (LCM) 200 mg given as 2 tablets of LCM 100 mg
Drug: Lacosamide (LCM) syrup — Treatment B: Single dose of Lacosamide (LCM) 200 mg given as syrup
  Arms: Treatment A - B

SUMMARY:
The purpose of this study is to demonstrate bioequivalence between the LCM tablet and syrup after single oral dosing in healthy Chinese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a Chinese male between 18 and 40 years of age
* Subject has no clinically significant cardiovascular, renal, gastrointestinal, hepatic, metabolic, endocrine, neurological, or psychiatric abnormalities and is in general good health
* Subject confirms that during the study and for a period of 3 months after the final dose of study drug, when having sexual intercourse with a woman of childbearing potential, an acceptable birth control method will be used

Exclusion Criteria:

Clinically significant

* out of range values for hematology and clinical chemistry variables
* abnormality in physical examination or vital signs
* ECG finding Any clinical conditions that in the opinion of the investigator would make the subject unsuitable for the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Lacosamide (LCM) | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Blood samples will be taken at indicated time points to determine maximum Lacosamide (LCM) plasma concentration.
Area under the LCM plasma concentration-time curve from time zero up to the time of last quantifiable concentration (AUC[0-t]) | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Area under the LCM plasma concentration-time curve from time zero up to the last quantifiable concentration data point, computed using the log-linear trapezoidal rule.
Area under the LCM plasma concentration-time curve extrapolated to infinity (AUC) | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Area under the LCM plasma concentration-time curve extrapolated to infinity calculated as AUC(0-t) + t/z, where t is the estimated plasma concentration at time t and z the terminal elimination rate constant.

SECONDARY OUTCOMES:
Terminal plasma elimination half-life (t1/2) of LCM | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Terminal elimination half-life of LCM, reported in hours, as determined via simple linear regression(slope=-z) of natural log (ln) concentration vs time for data points in the terminal phase of the concentration-time curve. t½ is calculated as ln(2)/z.
Time of observed Cmax (tmax) of LCM | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Time of observed Cmax will be obtained directly from the plasma concentration-time curves.
Apparent plasma clearance (CL/F) of LCM | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Apparent plasma clearance calculated as CL/F=Dose/AUC.
Apparent volume of distribution (Vz/F) of LCM | Blood samples are collected at predose and 0.25, 0.5, 1.0, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 72 hours after dosing
  Apparent volume of distribution, calculated as Vz/F=(CL/F)/z.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 877 822 9493)
Locations (1):
- Sp1001 001, Shanghai, China